CLINICAL TRIAL: NCT04560660
Title: Repeated Ketamine Treatment to Accelerate Efficacy of Prolonged Exposure in PTSD
Brief Title: Ketamine-enhanced Prolonged Exposure Therapy in PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-006-19F
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: PTSD
Keywords: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two parallel treatment conditions: 1) adjunctive ketamine infusions to prolonged exposure therapy or 2) adjunctive midazolam (active placebo) infusions to prolonged exposure therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators will use a sequentially numbered, opaque, sealed envelopes, pharmacy-controlled allocations, and coded identical containers for adequate concealment allocation. Administration of study drugs and infusion monitoring will be conducted by research nurse keeping blinding from investigators and independent outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine and prolonged exposure (PE) (Experimental): Single IV ketamine 0.5 mg/kg 24-72 hrs prior to PE session at week 1,2, and 3 followed by 7 additional PE sessions.
  Interventions: Drug: Ketamine
- Midazolam and prolonged exposure (PE) (Placebo Comparator): Single IV midazolam 0.045 mg/kg 24-72 hrs prior to PE session at week 1,2, and 3 followed by 7 additional PE sessions.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — FDA approved anesthetic medication with rapid acting antidepressant effects.
  Arms: Ketamine and prolonged exposure (PE)
Drug: Midazolam — FDA approved sedative medication with dissociative effects.
  Arms: Midazolam and prolonged exposure (PE)

SUMMARY:
The purpose of this study is to test the safety and efficacy of repeated doses of ketamine as compared to placebo to reduce symptoms of Posttraumatic Stress Disorder (PTSD) among Veteran receiving Prolonged Exposure Therapy.

DETAILED DESCRIPTION:
In this single site clinical trial, intended to evaluate the safety and efficacy of repeated doses of ketamine in conjunction with prolonged exposure (PE) therapy for PTSD. Veterans who meet criteria for PTSD and the additional inclusion and exclusion criteria will be randomized to one of two treatment arms (placebo plus PE vs ketamine plus PE). Participants receive the study drug via intravenous infusion once per week for 3-weeks.

ELIGIBILITY:
Inclusion Criteria:

* male or female Veterans between the ages of 18 and 75 years
* diagnosis of PTSD
* ability to provide written informed consent

Exclusion Criteria:

* females who are currently pregnant or breastfeeding
* current high risk for suicide
* history of moderate/severe head injury
* history of psychosis
* current episode of mania/hypomania
* severe substance and/or alcohol use disorder in the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | CAPS-5 to measure change in PTSD symptoms from baseline to post-treatment (10 weeks)
  The CAPS-5 is the gold standard in PTSD assessment consisting of a a 30-item structured interview. The CAPS-5 will be recorded and aggregated from all study participants. Range from 0 to 80 with higher score denoting more severe PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Shiroma, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04560660/ICF_000.pdf